CLINICAL TRIAL: NCT05377281
Title: Feasibility and Safety of autoloGous UncondItioneD pEripheral Nerve Tissue Delivery to the Substantia Nigra
Brief Title: Feasibility and Safety of autoloGous UncondItioneD pEripheral Nerve Tissue Delivery to the Substantia Nigra (GUIDE)
Acronym: GUIDE
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Craig van Horne, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Craig van Horne, MD, PhD, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 76436
Record Dates: First submitted 2022-05-04; First posted 2022-05-17 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Parkinson's Disease
Keywords: Peripheral nerve tissue
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implantation of peripheral nerve tissue (Experimental): Bilateral deployment of peripheral nerve tissue to the substantia nigra.
  Interventions: Procedure: Peripheral Nerve Tissue Implantation

INTERVENTIONS:
Procedure: Peripheral Nerve Tissue Implantation — At the time participants are receiving the standard of care deep brain stimulation (DBS) surgery, a standard incision on the lateral aspect near the ankle is made, the sural nerve is identified, an about 3 cm biopsy of the sural nerve is obtained and the incision is closed. From the biopsied section, the epineurium is removed, fascicles are cut, and (~5 pieces per side; ~ 5mm length x 1.5 mm diameter: approximately 10 cubic millimeters) implanted bilaterally into the substantia nigra.

SUMMARY:
This is an open-label, non-randomized, single-arm trial design to actively follow participants for 12 months. Ten participants will be enrolled to receive bilateral delivery of Peripheral Nerve Tissue (PNT) to the Substantia Nigra at the time of Deep Brain Stimulation (DBS) surgery. After 12 months, participants will be followed long term through annual visits for the rest of their lives. Participants will serve as their own donor for the tissue.

DETAILED DESCRIPTION:
We recently designed open-label safety studies to investigate the use of an autologous source of cellular tissue from the peripheral nervous system (van Horne et al., 2017, 2018; Quintero et al. 2022), reparative peripheral (sural) nerve tissue containing a variety of cells and neuroprotective factors (Chau et al. 2022). While our previous studies have used injury-activated peripheral nerve tissue (PNT), where the sural nerve is transected and allowed to regenerate in situ for up to about 2 weeks before implantation, here we propose to use naïve, previously uninjured, nerve tissue delivered bilaterally to the substantia nigra at the time participants are undergoing deep brain stimulation (DBS) surgery. Participants will be assessed preoperatively, then undergo DBS surgery and delivery of autologous PNT, and then assessed postoperatively at two weeks after surgery, 6 months, 12 months and annually thereafter for adverse events and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing DBS
* Diagnosis of clinically established or clinically probably PD (Parkinson's disease) as defined by MDS criteria
* Age 40-75, inclusive
* Able and willing to undergo ioflupane/SPECT
* Able to tolerate the surgical procedure
* Able to undergo all planned assessments
* Available access to the sural nerve

Exclusion Criteria:

* Any condition that would not make the subject a candidate for DBS
* Previous PD surgery or intracranial surgery
* Typical, nonparkinsonian syndrome ioflupane/SPECT signal
* Female who is pregnant, lactating, or of child-bearing potential unwilling to use an adequate birth control method during the period of the study
* Unable to undergo an MRI
* An obstructed trajectory path to the substantia nigra

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-07-07 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Implantation of peripheral nerve tissue (PNT) into the substantia nigra | 12 months
  Successful bilateral graft delivery to the substantia nigra at a proportion = 70%.

SECONDARY OUTCOMES:
Adverse Events | 12 months
  Number of adverse events and serious adverse events associated with bilateral PNT deployment to the substantia nigra.
Deployment | At the time of DBS surgery
  Number of deployment attempts required to deliver bilateral PNT
Procedure | At the time of DBS surgery
  Duration of procedure.
Admission | Surgery
  Length of hospital stay (days).
Retention | 12 months
  Percent of study visits completed.
Change in MDS-UPDRS scores | 12 months
  Mean change in MDS-UPDRS (Movement Disorder Society-Unified Parkinson's Disease Rating Scale) Part III scores for participants at 12, and 6 months compared to baseline.
  Mean change of the MDS-UPDRS Part I scores for participants at 6,12 months compared to baseline.
  Mean change of the MDS-UPDRS Part II scores for participants at 6,12 months compared to baseline. (95% confidence interval) Scale runs from 0-132 with smaller scores indicating fewer symptoms.
PDQ8 (Parkinson's Disease Questionnaire-8) | 12 months
  Mean change of the PDQ-8, Modified scores for participants at 6, 12 months compared to baseline. (95% confidence interval). Scale runs from 0-32 with lower scores indicating fewer symptoms.
Schwab and England | 12 months
  Mean change of the Modified Schwab and England Scale scores for participants at 6, 12 months compared to baseline. (95% confidence interval). Scale runs from 0%-100% with a higher score indicating the participant has more independence in their daily activities.
Neurocognitive Testing | 12 months post-surgery
  Mean change for neuropsychological assessment scores at 12 months compared to baseline. (95% confidence interval)

OTHER OUTCOMES:
Specific binding ratio | 12 months
  Mean change in specific binding ratio in the posterior putamen for participants at 12 months compared to baseline (95% confidence interval).

CONTACTS AND LOCATIONS:
Overall Officials: Craig van Horne, MD, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aparicio GI, Quintero JE, Plum L, Deng L, Wanczyk K, Henry M, Lynch E, Murphy M, Gerhardt GA, van Horne CG, Monje PV. Identification of cellular and noncellular components of mature intact human peripheral nerve. J Peripher Nerv Syst. 2024 Sep;29(3):294-314. doi: 10.1111/jns.12643. Epub 2024 Jul 7. PMID 38973168
- [Background] van Horne CG, Quintero JE, Slevin JT, Anderson-Mooney A, Gurwell JA, Welleford AS, Lamm JR, Wagner RP, Gerhardt GA. Peripheral nerve grafts implanted into the substantia nigra in patients with Parkinson's disease during deep brain stimulation surgery: 1-year follow-up study of safety, feasibility, and clinical outcome. J Neurosurg. 2018 Dec 1;129(6):1550-1561. doi: 10.3171/2017.8.JNS163222. Epub 2018 Feb 18. PMID 29451447
- [Background] Quintero JE, Slevin JT, Gurwell JA, McLouth CJ, El Khouli R, Chau MJ, Guduru Z, Gerhardt GA, van Horne CG. Direct delivery of an investigational cell therapy in patients with Parkinson's disease: an interim analysis of feasibility and safety of an open-label study using DBS-Plus clinical trial design. BMJ Neurol Open. 2022 Jul 14;4(2):e000301. doi: 10.1136/bmjno-2022-000301. eCollection 2022. PMID 35949912
- [Background] Quintero JE, Chau MJ, Slevin JT, Koehl L, Gurwell JA, Wallace E, Kryscio RJ, El Khouli R, Anderson-Mooney AJ, Schmitt FA, Gerhardt GA, van Horne CG. Two-year feasibility and safety of open-label autologous peripheral nerve tissue implantation during deep brain stimulation in patients with Parkinson's disease. J Parkinsons Dis. 2025 Mar;15(2):397-408. doi: 10.1177/1877718X241312409. Epub 2025 Feb 25. PMID 40007169